CLINICAL TRIAL: NCT00004312
Title: Establishment of a Database for Long-Term Monitoring of Patients With Nephropathic Cystinosis
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of California, San Diego (Other)
Other Study IDs: NCRR-M01RR00827-1196; UCSD-970026; UCSD-950338
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Cystinosis
Keywords: cystinosis; rare disease; renal and genitourinary disorders
MeSH Terms: conditions — Cystinosis; Rare Diseases; Urogenital Diseases

SUMMARY:
OBJECTIVES: I. Establish a computerized databank to monitor the progress of patients with cystinosis treated with cysteamine.

II. Track and monitor all patients including renal transplant, dialysis and post renal transplants.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Data are collected from patients and physicians. Information includes disease, treatment, family history, demographic, and physical exam data. The dates of kidney transplantation and/or dialysis initiation are also recorded.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

Nephropathic cystinosis diagnosis by white-cell cystine measurement, including infantile and late-onset forms

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Start 1999-10

CONTACTS AND LOCATIONS:
Overall Officials: Jerry A. Schneider, Study Chair — University of California, San Diego
Locations (1):
- University of California San Diego School of Medicine, La Jolla, California, United States